CLINICAL TRIAL: NCT00257075
Title: The Efficacy And Safety Of Flexible Dosage Ranges Of Risperidone Versus Placebo In The Treatment Of Manic Episodes Associated With Bipolar I Disorder.
Brief Title: A Study of the Effectiveness and Safety of Risperidone Versus Placebo in the Treatment of Manic Episodes Associated With Bipolar I Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR006052
Record Dates: First submitted 2005-11-18; First posted 2005-11-22 (Estimated); Last update posted 2011-01-14 (Estimated); Status verified 2011-01

CONDITIONS: Bipolar Disorders; Manic Episode
Keywords: risperidone; antipsychotic agents; bipolar disorders; manic episode
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — Risperidone

INTERVENTIONS:
Drug: Risperidone, oral tablets

SUMMARY:
The purpose of the study is to assess the effectiveness and safety of risperidone (an antipsychotic medication) versus placebo during 3 weeks of treatment of mania in patients with Bipolar I Disorder who are suffering a manic episode.

DETAILED DESCRIPTION:
Antipsychotic agents have, for a long time, been used to alleviate the severe behavioral problems associated with manic episodes. Risperidone, widely used in the treatment of schizophrenia, has been shown to be effective in the treatment of manic and mixed episodes associated with bipolar disorders. This is a randomized, double-blind, placebo-controlled study to evaluate the effectiveness and safety of risperidone compared with placebo in the treatment of patients with bipolar disorder who are experiencing a manic episode. Patients receive study medication (risperidone or placebo tablets) to be taken orally once a day at gradually increasing doses during the first week to achieve optimal effectiveness, while minimizing any intolerance to the drug. By Day 4, the dose of risperidone is in the range of 1 to 6 mg/day, and treatment with risperidone or placebo tablets continues for 3 weeks. The primary measure of effectiveness is the change in the Young Mania Rating Scale (YMRS) total score from baseline to the end of treatment. Additional assessments of effectiveness include the Clinical Global Impression-Severity of Illness (CGI-S) scale; the Global Assessment Scale (GAS), which assesses the patient's level of functioning; and the Positive and Negative Syndrome Scale (PANSS), a scale for measuring psychotic symptoms. Safety assessments include the incidence of adverse events throughout the study; measurement of vital signs (temperature, pulse, blood pressure) and evaluation of the presence and severity of extrapyramidal symptoms by the Extrapyramidal Symptom Rating Scale (ESRS) at specified intervals; and clinical laboratory tests (hematology, biochemistry, urinalysis) at the start and end of the study. The study hypothesis is that daily treatment with risperidone is more effective than placebo, as measured by Young Mania Rating Scale scores, in the treatment of the manic phase of Bipolar I Disorder. Risperidone tablets,1 mg (or placebo tablets) taken orally once daily in the evening; dose of 3 mg on Day 1; dose range of 2 - 4 mg on Day 2; dose range 1 - 5 mg on Day 3; dose range 1 - 6 mg on Days 4 - 21. Doses may be increased or decreased at investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of Bipolar I Disorder, Most Recent Episode Manic, by the criteria in the Diagnostic and Statistical Manual of Mental Diseases, 4th edition (DSM-IV)
* voluntarily hospitalized at study initiation for the current manic episode
* history of at least one documented manic or mixed episode that required treatment prior to study initiation
* total score of >=20 on the Young Mania Rating Scale (YMRS) and total score of <=20 on the Montgomery Asberg Depression Rating Scale (MADRS) at start of the study

Exclusion Criteria:

* Patients who meet DSM-IV criteria for Schizoaffective Disorder or for rapid cycling
* with borderline or antisocial personality disorder
* history of substance dependence (excluding nicotine and caffeine) within the 3 months prior to study initiation
* with seizure disorder
* females who are pregnant or nursing, or those lacking adequate contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2000-12; Study Completion 2002-05 (Actual)

PRIMARY OUTCOMES:
Change in Young Mania Rating Scale (YMRS) total score from baseline to the end of treatment.

SECONDARY OUTCOMES:
Change from baseline to the end of treatment in Clinical Global Impression-Severity of Illness (CGI-S) scale, Global Assessment Scale (GAS), and Positive and Negative Syndrome Scale (PANSS) total score; incidence of adverse events throughout study.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Hirschfeld RM, Keck PE Jr, Kramer M, Karcher K, Canuso C, Eerdekens M, Grossman F. Rapid antimanic effect of risperidone monotherapy: a 3-week multicenter, double-blind, placebo-controlled trial. Am J Psychiatry. 2004 Jun;161(6):1057-65. doi: 10.1176/appi.ajp.161.6.1057. PMID 15169694